CLINICAL TRIAL: NCT02472093
Title: A New Rehabilitation Tool in Fibromyalgia: Efficacy of Perceptive Rehabilitation Versus Group Exercises on Pain and Function: a Clinical Randomized Controlled Trial (RCT)
Brief Title: A New Rehabilitation Tool in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Teresa Paolucci, medical director, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2547-720/2012
Record Dates: First submitted 2015-06-06; First posted 2015-06-15 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2012-05

CONDITIONS: Fibromyalgia; Pain
Keywords: Postural exercise; Back pain; Tender points; Fibromyalgia; Perceptive rehabilitation
MeSH Terms: conditions — Fibromyalgia; Pain; Back Pain | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Physical exercises treatment (Active Comparator): The types of exercises included: low-impact to moderate aerobic training (gradually starting from 50% of the Fc max to 70%-80% of Fc max); walking fast in a circle, alternating with periods of going up and down the stairs (3 steps for 10 minutes) for a total of 20 consecutive minutes; posture exercises for the back and proprioceptive exercises for the trunk in the supine position to improve axial stability, including diaphragmatic breathing.
  Interventions: Other: Physical exercises treatment
- Perceptive Rehabilitation Treatment (Experimental): Perceptual surfaces is a therapeutic system that is based on the interaction between the patient's back or painful area and a support surface, composed of small latex cones with various dimensions (height: 3-8 cm; base diameter: 2-4 cm) and elasticities. The inferior bases of these cones are applied to a rigid wood surface using elastic strips; usually, over 100 cones are used for each session. Patients were asked to lie down supine on the surface that was formed by the smoothed apex of these cones, creating reaction forces to the patient's weight, generated by the interaction with the cones.
  Interventions: Other: Perceptive Rehabilitation Treatment
- Control group (Active Comparator): The control group did brief educational sessions.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Physical exercises treatment — Includes different types of exercises: low-impact to moderate aerobic training; walking fast in a circle, alternating with periods of going up and down the stairs (3 steps for 10 minutes) for a total of 20 consecutive minutes; posture exercises for the back and proprioceptive exercises for the trunk in the supine position to improve axial stability, including diaphragmatic breathing. The heart rate was monitored through the use of a heart rate monitor, which allowed not to exceed the threshold.
  Other Names: Rehabilitation Group Exercises
  Arms: Physical exercises treatment
Other: Perceptive Rehabilitation Treatment — therapeutic system that is based on the interaction between the patient's back or painful area and a support surface, composed of small latex cones with various dimensions (height: 3-8 cm; base diameter: 2-4 cm) and elasticities. The inferior bases of these cones are applied to a rigid wood surface using elastic strips.
  Other Names: Perceptual surfaces
  Arms: Perceptive Rehabilitation Treatment
Other: Control group — The control group did brief educational sessions.
  Arms: Control group

SUMMARY:
The aim of the investigators study was to measure reductions in chronic pain in female patients with Fibromylgia comparing individual proprioceptive rehabilitation treatments with perceptual surfaces to a group exercises rehabilitation. Fibromyalgia is a generalized chronic pain condition that is usually accompanied by fatigue, sleep disturbance and psychological and cognitive alterations.

ELIGIBILITY:
Inclusion Criteria:

* fibromyalgia diagnosed according to the criteria proposed by the American College of Rheumatology (ACR 1990 and 2010)
* Subjects aged between 18 and 60 years
* visual analog scale (VAS) for pain > 5

Exclusion Criteria:

* presence of concomitant autoimmune diseases
* psychiatric disorders
* other causes of chronic pain
* other diseases that prevented physical loading
* severe scoliosis or kyphoscoliosis
* surgery of the spine
* vertebral fractures
* sciatic pain
* tumors
* enrolled in another type of physical therapy program
* myocardial infarction
* lower extremity arterial disease
* major neurological problems
* diabetes
* gastrointestinal disease
* chronic respiratory disease
* kidney disease
* poor vision

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change of Fibromyalgia Assessment Scale (FAS) from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  It is a simple and rapidly implemented index, consisting of a pain map, called the Self-Assessment Pain Scale (SAPS) (in which the patient is asked to indicate how much pain he suffered in the previous week in 16 areas of the body, with scored from 0 to 3), and 2 scales (between 0 and 10) that evaluate fatigue and quality of sleep, scored from 0-10. The FAS allows physicians to obtain reliable information concerning the course of the disease and is sufficiently sensitive to alert them in case of deterioration.

SECONDARY OUTCOMES:
Change of Fibromyalgia Impact Questionnaire (FIQ) from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  It comprises 3 sections-function, impact, and symptoms-combining to generate an overall score. The first section contains 10 sub items and focuses on the patient's ability to perform daily tasks that involve the large muscles (eg, cooking, cleaning, walking, shopping, homemaking, socializing, and mobility). The next 2 items ask patients to circle the number of days in the past week in which they felt good and the number of days that they missed work. The last 7 items assess the ability to do one's job, pain, fatigue, morning tiredness, stiffness, anxiety, and depression. The total score on the FIQ is calculated by adding the following 10 items: the physical function score, the number of days feeling good, the number of work days missed, the ability to do one's job, pain, fatigue, morning tiredness, stiffness, anxiety, and depression. The FIQ score ranges from 0 to 100, with 100 indicating the worst possible score due to Fibromylgia.
Change of Health Assessment Questionnaire (HAQ) from baseline to 12 weeks | baseline, 4 weeks, 12 weeks
  It is a 20-item self-administered questionnaire that determines the difficulty in performing 8 daily activities (dressing and grooming, getting up, eating, walking, hygiene, reaching, ability to grip, and outside activities). For each item, patients are asked to rate the level of difficulty that they have experienced over the previous week in performing these activities on a 4-point scale from 0 (no difficulty) to 3 (unable to perform). The final HAQ score is the average score of the 8 categories, thus ranging from 0 to 3; higher scores reflect greater levels of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Maria Saraceni, Principal Investigator — Umberto I Hospital, Sapienza University of Rome